CLINICAL TRIAL: NCT00646984
Title: Comparison of Strategies of Interruption/Reinitiation of Antiretroviral Therapy in Response to Immunologic/Virologic Changes in HIV-Infected Patients With Lipodystrophy.
Brief Title: Strategies of Interruption/Reinitiation of Antiretroviral Therapy in HIV-Infected Patients With Lipodystrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Esteban Martinez, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TARV-DEM-LD; AEM 01-0480
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: HIV-Associated Lipodystrophy Syndrome
Keywords: Lipodystrophy; Treatment interruption; HIV
MeSH Terms: conditions — HIV-Associated Lipodystrophy Syndrome; Lipodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Standard continuous antiretroviral therapy
  Interventions: Drug: Standard continuous antiretroviral therapy
- 2 (Experimental): CD-4 guided interruption arm
  Interventions: Drug: CD-4 guided therapy interruption
- 3 (Experimental): Viral load driven treatment interruption
  Interventions: Drug: Viral load driven treatment interruption

INTERVENTIONS:
Drug: Standard continuous antiretroviral therapy
  Arms: 1
Drug: CD-4 guided therapy interruption — Stop antiretroviral therapy when CD-4 equal or above 350 and reinitiate when below 350
  Arms: 2
Drug: Viral load driven treatment interruption — Stop antiretroviral therapy when viral load below 30,000 copies/ml and reinitiate when equal or above 30,000 copies/ml
  Arms: 3

SUMMARY:
Aim: To assess the safety on the progression of HIV infection and the efficacy on the evolution of metabolic parameters and body fat of either viral load- or CD4 cell-driven strategies of intermittent treatment in chronically HIV-1-infected persons.

Design: Pilot, prospective, open, randomized, controlled 3-year study.

Setting and patients: University hospital. Patients with viral load <200 copies/mL and CD4 cell count >450/mm3 for at least the last 3 months. Three arms with 50 patients each, that will be randomized either to continue antiretroviral therapy, or to discontinue it as long as either HIV-1 RNA be lower than 30000 copies/mL or CD4 cell count be higher than 300/mm3.

Study end-points: evolution of plasma metabolic parameters, body fat, and bone mineral density; incidence of adverse effects due to antiretroviral therapy and symptoms consistent with acute retroviral syndrome; incidence of virological failure (plasma HIV-1 RNA >200 copies/mL while on therapy), immunological failure (CD4 cell count <200/mm3 while on therapy), or clinical failure (development of AIDS-defining illnesses); cost of antiretroviral therapy administered and time free of therapy in the arms assigned to intermittent treatment; and the evolution of T lymphocyte subpopulations and the development of proliferative and cytotoxic responses against HIV.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients
* On stable antiretroviral therapy
* Viral load below 200 copies/ml
* CD4 above 450 cells/mcl during last 3 months

Exclusion Criteria:

* Weight variation higher than 10% compared with previous stable weight
* Active (CDC-C) opportunistic events
* Major depression or schizophrenia under psychiatric treatment
* Lack of clinical stability
* Pregnant women or planning pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2002-01; Primary Completion 2005-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Limb fat content measured by dual X-ray absorptiometry | 96 weekks

SECONDARY OUTCOMES:
Other body composition analyses | 96 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Gatell, MD, Study Director — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain